CLINICAL TRIAL: NCT00939575
Title: Feasibility Study to Develop Analysis of the Metabolomics Patterns of Women With Hypertensive Disorders During Pregnancy.
Brief Title: Pre-eclampsia and Metabolomics
Acronym: GEM-1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Foundation of the Stars (Other)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, Pr, Université de Sherbrooke
Other Study IDs: 08-173
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Preeclampsia
Keywords: preeclampsia, metabolomics, blood, urine
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and urine are collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preeclampsia: Women hospitalized for pre-eclampsia after 20 0/7 weeks of gestation. The diagnosis of preeclampsia include a combination of the following criteria: after 20 weeks of gestation in a previously normotensive woman, a diastolic blood pressure > 90 mmHg recorded twice at least four hours apart or > 110 mmHg, with proteinuria > 300 mg/24h or > 30 mg / mmol protein / urinary creatinine in a urine sample or factor (s) serious maternal / fetal (according to SOGC consensus ).
- control: Women will be matched to women with pre-eclampsia according to gestational age at diagnosis of preeclampsia, maternal age (in stratum of 5 years), gender, ethnicity (4 categories: Caucasian, black, Asian and other) and body mass index (5 classes: <20, 20-25, 26-30, 31-35 and <35). Patients of this group should be at low risk of obstetric complications at recruitment and planning to deliver at the CHUS.

SUMMARY:
The hypertensive disorders of pregnancy are the medical complications more prevalent during pregnancy. In Canada, approximately 1% of pregnancies have complications due to a pre-existing hypertension, 5-6% because of hypertension of pregnancy without proteinuria and 1-2% by preeclampsia. Metabolomics involves a new technology to investigate small molecules that characterize biochemical pathways of interest. The change in concentration levels of these molecules in various biological samples such as urine and blood in the presence of a disease or a patient can be particularly useful for identifying new biomarkers. Our hypothesis is that metabolic patterns in blood and urine of pregnant women who had preeclampsia differ from the metabolomics patterns of patients without preeclampsia.The whole research program has two complementary objectives in order to expect a decrease of prematurity: a) better understanding of all the physiological mechanisms leading to prematurity and b) better identification of patients at high risk for a better management of these women.

DETAILED DESCRIPTION:
Metabolomics involves a new technology using the methods of separation and detection complex to investigate a set of small molecules that characterize biochemical pathways of interest. The change in concentration levels of these molecules in various biological samples such as urine and blood in the presence of a disease or a patient can detect metabolic fingerprints that can be particularly useful for identifying new biomarkers. These will thereafter be quantified and validated by metabolic profiling. To our knowledge, there are few studies on metabolomics and pregnancy.

Methods:

The studied population will be women hospitalized for preeclampsia (after 20 SA). Women in the control group will be matched to women hospitalized for pre-eclampsia according to gestational age at diagnosis of pre-eclampsia, maternal age, parity, ethnicity and body mass index.

Blood and urine samples will be taken:

Case control:

* Following the diagnosis of preeclampsia
* At each blood test requested by the physician during the follow-up
* When the patient will be in labor (cervix ripening > 5 cm) or before the caesarean section
* 48 hours after delivery
* 6-8 weeks after delivery

Control group:

* Following the inclusion as a control in the study
* At admission for delivery
* When the patient will be in labor (dilation > 5 cm) or before the caesarean section
* 48 hours after delivery
* 6-8 weeks after delivery

ELIGIBILITY:
Inclusion Criteria:

* Case group: Women hospitalized for pre-eclampsia after 20 0/7 weeks of gestation. The diagnosis of preeclampsia include a combination of the following criteria: after 20 weeks of pregnancy in a previously normotensive woman, a diastolic blood pressure ≥ 90 mmHg recorded twice at least four hours apart or ≥ 110 mmHg, with proteinuria ≥ 300 mg/24h or ≥ 30 mg / mmol protein / urinary creatinine in a urine sample or factor (s) serious maternal / fetal (according to consensus SOGC).
* Control group: Women will be matched to women with preeclampsia according to gestational age at diagnosis of pre-eclampsia, maternal age (in stratum of 5 years), gender, ethnicity (4 categories: Caucasian, black, Asian and other) and body mass index (5 classes: < 20, 20-25, 26-30, 31-35 and < 35). Patients of this group should be at low risk of obstetric complications at recruitment and planning to deliver at the CHUS.

Exclusion Criteria:

- Minor patients, patients with post-partum preeclampsia, premature rupture of membranes, a severe congenital fetal malformation, twin pregnancies and fetal death. Patients with underlying diseases taht could be associated with preeclampsia as pre-existing hypertension (ie before 20SA), anti-phospholipid syndrome, lupus, type DM 1-2, nephropathy, etc will be excluded. Patients who have a complication during the pregnancy will be excluded from the control group.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women who deliver at the CHUS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
comparison between the metabolic patterns of women hospitalized for preeclampsia and the control group | between diagnosis of preeclampsia (or equivalent gestational age) and delivery

SECONDARY OUTCOMES:
Longitudinal comparison of metabolomics patterns of the same individual | between diagnosis of preeclampsia and 2 months after delivery
Compare metabolomics patterns of pregnant women with preeclampsia early (<34 weeks) during pregnancy to those women with pre-eclampsia later during pregnancy (≥34 weeks of gestation). | between diagnosis of preeclampsia and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Sherbrooke; Christiane Auray-Blais, PhD, Principal Investigator — Centre hospitalier de l'Université de Sherbrooke
Locations (1):
- Centre hospitalier de l'Université de Sherbrooke, Sherbrooke, Quebec, Canada